CLINICAL TRIAL: NCT00416091
Title: Neuropsychological Functioning, Symptomatology, and Social Adjustment Among Children With Tourret's Disorder, Attention-Deficit/Hyperactivity Disorder, and Comorbid Conditions.
Brief Title: Neuropsychological Functioning Among Children With Tourret's Disorder and ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9561706006; NTUH96- S558 (Other: National Taiwan University Hospital)
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2008-09

CONDITIONS: Tourette Disorder; Attention-Deficit/Hyperactivity Disorder
Keywords: Tourette disorder, ADHD, comorbidity, neuropsychological
MeSH Terms: conditions — Tourette Syndrome; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tourette's disorder (TD) is a childhood-onset neuropsychiatric disorder, manifesting motor and vocal tics with increased likelihood of comorbid with attention-deficit/hyperactivity disorder (ADHD) and other psychiatric disorders. Literature documents the comorbid condition with ADHD predicts an increased functional deficit among individuals with ADHD. The information about neuropsychological functioning among individuals with TD adn/or ADHD is little in Asian population. This study aims to validate the diagnoses of TD, ADHD, and TD comorbid ADHD by symptomatology, neuropsychological measures, and social adjustment. This is a case-control study with a sample of 30 subjects with TD, 60 with ADHD, 30 with TD+ADHD, and 60 controls aged from 6 to 18. All subjects will receive comprehensive assessment including standard psychiatric diagnostic interviews using (K-SADS-E), behavioral assessments (SNAP-IV, CPRS:R-S, CTRS:R-S, CBCL, YBOCS, YGTSS), social adjustment (SAICA, GCAS), parenting (PBI, APGAR) and neuropsychological assessment (CPT, CANTAB, WISC-III). We anticipate that this study will provide the primitive data to validate the TD and ADHD using neuropsychological and clinical measures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 8-16 without the diagnosis of ADHD, and/or Tourette's disorder
* IQ > 80
* both children/adolescents and their parents consent to participate and have the ability to complete self-administered measures in this study

Exclusion Criteria:

* diagnosis of psychotic disorders, bipolar affective disorders, pervasive developmental disorder, seizure, or major physical disorders.
* in addition, control subjects will be excluded from the control group if have a history of the following condition as defined by DSM-IV: ADHD, ODD, or CD in addition to the above exclusion criteria.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ADHD, children with ADHD and Tourette's disorder, normal control
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Barkley RA (1997), Behavioral inhibition, sustained attention, and executive functions: constructing a unifying theory of ADHD. Psychol Bull 121: 65-94 Channon S, Pratt P, Robertson MM (2003b), Executive function, memory, and learning in Tourette's disorder. Neuropsychology 17: 247-54 Gau SS, Soong WT, Chiu YN, Tsai WC (2006a), Psychometric properties of the Chinese version of the Conners' Teacher and Parent Rating Scales-Revised Short Form. Journal of Attention Disorders. 9: 648-659 Gau SSF, Shen HY, Soong WT, Gau CS (2006b), An open-label, randomized, active controlled equivalent trial of OROS methylphenidate in children with attention-deficit/hyperactivity disorder in Taiwan. Journal of Child and Adolescent Psychopharmacology 16 (in press) Kurlan R, Whitmore D, Irvine C, McDermott MP, Como PG (1994), Tourette's disorder in a special education population: a pilot study involving a single school district. Neurology 44: 699-702